CLINICAL TRIAL: NCT06602973
Title: Relationships Between Exercise and Appetite in Women With Loss of Control Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Katherine J. Forney, Assistant Professor, Ohio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_FY24-403
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders; Binge-Eating Disorder; Bulimia Nervosa
Keywords: exercise; eating disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Bulimia Nervosa; Motor Activity | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Rest, Fed Exercise, Fasted Exercise (Experimental): At Study Visit 2, participants will eat breakfast and rest (abstain from exercise).
  At Study Visit 3, participants will eat breakfast and exercise. At Study Visit 4, participants will abstain from breakfast and will engage in exercise.
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise
- Rest, Fasted Exercise, Fed Exercise (Experimental): At Study Visit 2, participants will eat breakfast and rest (abstain from exercise).
  At Study Visit 3, participants will abstain from breakfast and will engage in exercise.
  At Study Visit 4, participants will eat breakfast and exercise.
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise
- Fed Exercise, Rest, Fasted Exercise (Experimental): At Study Visit 2, participants will eat breakfast and exercise. At Study Visit 3, participants will eat breakfast and rest (abstain from exercise).
  At Study Visit 4, participants will abstain from breakfast and will engage in exercise.
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise
- Fed Exercise, Fasted Exercise, Rest (Experimental): At Study Visit 2, participants will eat breakfast and exercise. At Study Visit 3, participants will abstain from breakfast and will engage in exercise.
  At Study Visit 4, participants will eat breakfast and rest (abstain from exercise).
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise
- Fasted Exercise, Fed Exercise, Rest (Experimental): At Study Visit 2, participants will abstain from breakfast and will engage in exercise.
  At Study Visit 3, participants will eat breakfast and exercise. At Study Visit 4, participants will eat breakfast and rest (abstain from exercise)
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise
- Fasted Exercise, Rest, Fed Exercise (Experimental): At Study Visit 2, participants will abstain from breakfast and will engage in exercise.
  At Study Visit 3, participants will eat breakfast and rest (abstain from exercise).
  At Study Visit 4, participants will eat breakfast and exercise.
  Interventions: Behavioral: Rest; Behavioral: Fed Exercise; Behavioral: Fasted Exercise

INTERVENTIONS:
Behavioral: Rest — Participants will eat breakfast but abstain from exercise
Behavioral: Fed Exercise — Participants will eat breakfast and engage in 30 minutes of physical activity at 75% of their personal V02max.
Behavioral: Fasted Exercise — Participants will engage in 30 minutes of physical activity at their personal 75% V02max after abstaining from breakfast.

SUMMARY:
This pilot study is a first step in looking at the relationship between exercise and appetite in women with loss of control eating.

ELIGIBILITY:
Inclusion Criteria:

* Engage in loss of control eating at least 12 times in the last three months
* Clinically significant eating disorder-related impairment (CIA > 15)
* Taking hormonal contraception
* Minimum VO2max of 50th percentile for age and sex assigned at birth
* Be willing to eat study-provided foods
* Likes chocolate (at least 6/10 on 10 point scale)

Exclusion Criteria:

* BMI < 18.5 kgm/2
* Medical conditions that affect appetite or weight (e.g., diabetes mellitus, thyroid disease)
* Recent pregnancy or breastfeeding (prior 6 months)
* Relevant food allergies (e.g., wheat, chocolate)
* Specific phobia, blood-injection-injury type
* Medical condition that precludes safe participation in exercise (e.g., stress fracture)
* Medications that acutely affect appetite (e.g., GLP-1 agonists; psychiatric medications allowed)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Relative Energy Intake | Food intake from 8 am to 8 am; Energy expenditure from approximately 9 am to 9:05 am and 9:25 to 9:30 am, coinciding with study condition (rest or exercise)
  Relative energy intake for 24 hours will be calculated as absolute energy intake from the breakfast (if consumed), lunch, food reward value task, and take home cooler minus energy expenditure during exercise (or comparable time period during rest).

SECONDARY OUTCOMES:
Lactate | 30 minutes, pre-post exercise (or rest)
  Lactate values
Acylated ghrelin | Immediately prior to lunch
  Acylated ghrelin
Self-reported binge eating | 24 and 48 hours after exercise/rest study visit
  Participants will rate the extent the following questions, considering the time frame "since yesterday morning at 8 am" on a 1 to 5 scale from "not at all" to "extremely":
  "While you were eating, to what extent did you feel a sense of loss of control?," "While you were eating, to what extent did you feel that you could not resist eating," "While you were eating, to what extent did you feel that you could not stop eating once you had started," and "While you were eating, to what extent did you feel driven or compelled to eat?" An answer of 4 or higher on any item will be categorized as binge eating present. Any reported binge eating on either day will be coded as binge eating being present
Food reward value | Approximately 3:30 pm day of study visit
  Number of trials according to task developed by Bodell and Keel 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared on a public repository, such as the Open Science Framework